CLINICAL TRIAL: NCT05405192
Title: Phase 2 Single Agent Dostarlimab in Chemoresistant Gestational Trophoblastic Neoplasia (GTN)
Brief Title: Dostarlimab in Chemoresistant Gestational Trophoblastic Neoplasia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI is leaving the University.
Sponsor: University of Miami (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20210967
Record Dates: First submitted 2022-05-26; First posted 2022-06-06 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Gestational Trophoblastic Neoplasia
MeSH Terms: conditions — Gestational Trophoblastic Disease | interventions — dostarlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dostarlimab Group (Experimental): Participants will receive a total of up to 20 cycles of Dostarlimab: 4 cycles of Dostarlimab at a dose of 500 mg on day 1 of each of the 21-day cycle and 16 cycles of Dostarlimab at a dose of 1000 mg on day 1 of each of the 42-day cycle.
  Interventions: Drug: Dostarlimab

INTERVENTIONS:
Drug: Dostarlimab — First four cycles of Dostarlimab will be given intravenously (IV) on day 1 of each of the 21-day cycle at a dose of 500 milligrams (mg). The next 16 cycles of Dostarlimab will be given on day 1 of each of the 42-day cycles at a dose of 1,000 mg.

SUMMARY:
The purpose of this study is to see if Dostarlimab is an effective treatment for Gestational Trophoblastic Neoplasia (GTN).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with persistent unresectable Gestational Trophoblastic Neoplasia (GTN) disease
2. Female patients >18 years old.
3. Pretreatment archival tissue (if available) must be submitted for correlative studies. If pre-treatment tissue is not available, this does not exclude the patient.
4. Patients must have recovered from the effects of recent surgery or radiotherapy (persistent toxicity, CTCAE grade ≤1 except for alopecia, sensory neuropathy, or fatigue).

Exclusion Criteria:

1. Prior therapy with anti-Programed Death (PD)1/Programed Death Ligand-1 (PD-L1) or anti-CTLA4 antibody
2. Participant must not be simultaneously enrolled in any interventional clinical trial.
3. Participant must not have had major surgery ≤3 weeks prior to initiating protocol therapy and participant must have recovered from any surgical effects.
4. Participant must not have received investigational therapy ≤ 4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is shorter, prior initiating protocol therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with successful normalization of beta hCG | Up to 24 months
  Proportion of patients with a successful normalized serum human chorionic gonadotropin (hCG) level (complete response) as measured by serum samples.

SECONDARY OUTCOMES:
Proportion of patients with objective response rate (ORR) | Up to 25 months
  ORR is defined as achieving best response of complete or partial responses (CR or PR) as assessed via Response Evaluated Criteria in Solid Tumors (RECIST)
Number of Participants with treatment related-adverse events | Up to 25 months
  Non-hematological Grade 3 and higher treatment-related adverse events as evaluated by treating physician using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.
Progression-free survival (PFS) | Up to 48 months
  PFS is the elapsed time from the date of treatment initiation to date of first documentation of progression (or recurrence) or death due to any cause. Patients last known to be alive and free of disease will be censored at date of last documented progression-free status.
Overall survival (OS) | Up to 48 months
  OS is the elapsed time from treatment initiation to death. For alive patients, OS will be censored at the date last known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Huang, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No